CLINICAL TRIAL: NCT06493344
Title: The Influence of Applying Additional Weight on Crouch Gait in Children With Spastic Cerebral Palsy. Assessment of the Kinematics, Balance and Functional Level
Brief Title: The Influence of Applying Additional Weight on Crouch Gait in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, George Paras, Assistant Professor, University of Thessaly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: add-weight-CP
Record Dates: First submitted 2024-06-26; First posted 2024-07-10 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy; Gait, Spastic; Motor Disorders; Functional Neurological Disorder
Keywords: cerebral palsy; crouch gait; physiotherapy; balance; kinematic analysis
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic; Motor Disorders; Conversion Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spastic Cerebral Palsy Group (Experimental): Conventional physiotherapy and training with applying additional weight
  Interventions: Other: Applying additional weight

INTERVENTIONS:
Other: Applying additional weight — Treadmill training with and without weight (15 minutes of 3 times/ per week for 16 weeks).

SUMMARY:
The purpose of this study was to investigate the effectiveness of applying additional weight in the improvement of the crouch gait pattern in children with spastic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

The children who participated in the study, aged 12 - 15 years old, were diagnosed with spastic cerebral palsy, level III according to the classification of the GMFCS.

Exclusion Criteria:

From the study, they were excluded:

1. children who have received botulinum toxin injection up to 3 months before,
2. children who have had selective rhizotomy surgery up to 1 year before,
3. children who have a baclofen pump,
4. children with uncontrolled epilepsy,
5. children with cognitive deficits who cannot follow verbal instructions.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Kinovea | up to 16 weeks (every 4 weeks)
  Kinovea is a 2D video annotation tool designed for kinematic analysis. Assessment of knee angle during stance phase.
Gross Motor Function Measure 88 (GMFM-88) | up to 16 weeks (every 4 weeks)
  An assessment tool designed and evaluated to measure changes in gross motor function over time in children with cerebral palsy. Unit of Measure: Scoring Options (0, 1, 2, 3, or "not tested") // (higher scores - better outcome)
Timed Up and Go | up to 16 weeks (every 4 weeks)
  The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk in disabled children. Unit of measure: seconds of completion (higher scores - worse outcomes)
Sit to Stand (STS) test of the NeuroCom® Balance Master® | up to 16 weeks (every 4 weeks)
  A cutting-edge technology used at Balance and Mobility Therapy to accurately assess and treat balance disorders.

CONTACTS AND LOCATIONS:
Overall Officials: George Paras, Ph.D., Principal Investigator — University of Thessaly
Locations (1):
- Department of Physiotherapy - University of Thessaly, Lamia, Phthiotis, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verschuren O, Peterson MD, Balemans AC, Hurvitz EA. Exercise and physical activity recommendations for people with cerebral palsy. Dev Med Child Neurol. 2016 Aug;58(8):798-808. doi: 10.1111/dmcn.13053. Epub 2016 Feb 7. PMID 26853808
- [Background] Merino-Andres J, Garcia de Mateos-Lopez A, Damiano DL, Sanchez-Sierra A. Effect of muscle strength training in children and adolescents with spastic cerebral palsy: A systematic review and meta-analysis. Clin Rehabil. 2022 Jan;36(1):4-14. doi: 10.1177/02692155211040199. Epub 2021 Aug 18. PMID 34407619